CLINICAL TRIAL: NCT07362979
Title: Toripalimab Combined With Different Platinum-Based Induction Chemotherapy Regimens for Locally Advanced Nasopharyngeal Carcinoma: A Randomized, Open-label, Controlled, Multicenter Phase II Trial
Brief Title: Toripalimab Combined With Different Platinum-Based Induction Chemotherapy Regimens for Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-446
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; Toripalimab; different platinum-based induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — CCDC6 protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GP plus Toripalimab Induction chemotherapy (Experimental): Induction Chemotherapy + Immunotherapy (3 Cycles): Gemcitabine 1000mg/m^2 (Days 1, 8) + Cisplatin 80mg/m^2 (Day 1) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles.
  Interventions: Drug: GP plus Toripalimab Induction chemotherapy+CCRT
- TP plus Toripalimab Induction chemotherapy (Experimental): Induction Chemotherapy + Immunotherapy (3 Cycles): Nab-paclitaxel 260mg/m^2 (Days 1) + Cisplatin 75mg/m^2 (Day 1) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles.
  Interventions: Drug: TP plus Toripalimab Induction chemotherapy+CCRT
- TPC plus Toripalimab Induction chemotherapy (Experimental): Induction Chemotherapy + Immunotherapy (3 Cycles): Nab-paclitaxel 200mg/m^2 (Days 1) + Cisplatin 75mg/m^2 (Day 1) + Capecitabine 1000mg/m^2 BID (Day 1-Day14) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles.
  Interventions: Drug: TPC plus Toripalimab Induction chemotherapy+CCRT

INTERVENTIONS:
Drug: GP plus Toripalimab Induction chemotherapy+CCRT — Induction Chemotherapy + Immunotherapy (3 Cycles):
  Gemcitabine 1000mg/m^2 (Days 1, 8) + Cisplatin 80mg/m^2 (Day 1) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles. Sequentially followed by Concurrent Chemoradiotherapy (CCRT): Cisplatin 100mg/m^2 (Day 1), administered every 3 weeks for a total of 3 cycles during the radiotherapy period (on Days 1, 22, and 43 of radiotherapy).
  Arms: GP plus Toripalimab Induction chemotherapy
Drug: TP plus Toripalimab Induction chemotherapy+CCRT — Induction Chemotherapy + Immunotherapy (3 Cycles):
  Nab-paclitaxel 260mg/m^2 (Days 1) + Cisplatin 75mg/m^2 (Day 1) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles. Sequentially followed by Concurrent Chemoradiotherapy (CCRT): Cisplatin 100mg/m^2 (Day 1), administered every 3 weeks for a total of 3 cycles during the radiotherapy period (on Days 1, 22, and 43 of radiotherapy).
  Arms: TP plus Toripalimab Induction chemotherapy
Drug: TPC plus Toripalimab Induction chemotherapy+CCRT — Induction Chemotherapy + Immunotherapy (3 Cycles):
  Nab-paclitaxel 200mg/m^2 (Days 1) + Cisplatin 75mg/m^2 (Day 1) + Capecitabine 1000mg/m^2 BID (Day 1-Day14) + Toripalimab 240mg (Day 1), administered every 3 weeks for a total of 3 cycles. Sequentially followed by Concurrent Chemoradiotherapy (CCRT): Cisplatin 100mg/m^2 (Day 1), administered every 3 weeks for a total of 3 cycles during the radiotherapy period (on Days 1, 22, and 43 of radiotherapy).
  Arms: TPC plus Toripalimab Induction chemotherapy

SUMMARY:
This phase II randomized trial compares the efficacy and safety of Toripalimab combined with three different platinum-based induction chemotherapy regimens, sequentially followed by standard concurrent chemoradiotherapy, for the treatment of locally advanced nasopharyngeal carcinoma (NPC). The study is aimed to pick up the most effective platinum-based induction chemotherapy regimen plus Toripalimab for these patients which provides the most survival benefit.

DETAILED DESCRIPTION:
This phase II randomized trial compares the efficacy and safety of Toripalimab combined with three different platinum-based induction chemotherapy regimens, sequentially followed by standard concurrent chemoradiotherapy, for the treatment of locally advanced nasopharyngeal carcinoma (NPC). The enrolled patients will be 1:1:1 randomly assigned to receive induction chemotherapy of Gemcitabine plus Cisplatin plus Toripalimab(GP plus Toripalimab regimen), Nab-paclitaxel plus Cisplatin plus Toripalimab (TP plus Toripalimab regimen) or Nab-paclitaxel plus Cisplatin plus Capecitabine plus Toripalimab(TPC plus Toripalimab regimen).The study is aimed to pick up the most effective platinum-based induction chemotherapy regimen plus Toripalimab for these patients which provides the most survival benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years, male or non-pregnant female.
2. Pathologically confirmed nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
3. Stage Any T, N2-3 or T4, N1 (AJCC 9th edition staging), with no distant metastasis (M0).
4. ECOG performance status score of 0 or 1.
5. Adequate hematological function: Hemoglobin (HGB)≥90g/L, Absolute Neutrophil Count (ANC) ≥ 1.5*10^9/L, and Platele (PLT) ≥100*10^9/L.
6. Adequate hepatic function: ALT and AST≤2.5*Upper Limit of Normal (ULN), total bilirubin ≤2.0*ULN, and serum albumin≥30g/L.
7. Adequate renal function: Serum creatinine ≤ 1.5*ULN or calculated creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault formula).
8. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 *ULN (unless the subject is receiving anticoagulant therapy and the coagulation parameters (PT/INR and APTT) are within the expected therapeutic range for the anticoagulant at the time of screening).

Exclusion Criteria:

1. Patients with nasopharyngeal carcinoma presenting with recurrence or distant metastasis.
2. Pathologically confirmed diagnosis of keratinizing squamous cell carcinoma (WHO Type I).
3. Prior history of radiotherapy or systemic chemotherapy.
4. Women who are pregnant, lactating, or of childbearing potential not employing effective contraception.
5. HIV-positive status.
6. History of other malignancies (except for cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Patients previously treated with immune checkpoint inhibitors (e.g., CTLA-4, PD-1, PD-L1 inhibitors).
8. Patients with immunodeficiency diseases or a history of organ transplantation.
9. Patients who have received high-dose glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressive therapy within 4 weeks prior.
10. Patients with significantly impaired cardiac, hepatic, pulmonary, renal, or bone marrow function.
11. Concurrent use of other investigational drugs or current participation in another clinical trial.
12. Patients who refuse or are unable to provide signed informed consent for trial participation.
13. Patients with personality or psychiatric disorders, or those lacking legal capacity or with limited legal capacity.
14. Hepatitis B surface antigen (HBsAg) positive with peripheral blood Hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 1000 copies/ml.
15. Patients with positive Hepatitis C virus (HCV) antibody test results are eligible only if the HCV ribonucleic acid (RNA) polymerase chain reaction test result is negative.
16. Arterial or venous thrombotic events within 6 months prior to screening initiation, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism.
17. Known history of active tuberculosis (TB). Subjects suspected of having active TB must be evaluated and ruled out via chest X-ray, sputum examination, and clinical signs and symptoms.

21.Any other severe, uncontrolled medical condition, infection, or treatment contraindication, or any other condition that, in the investigator's judgment, may pose a risk for receiving the investigational drug, or may interfere with the assessment of the investigational drug, subject safety, or interpretation of the study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2031-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The time from randomization to any documented local or regional relapse, distant metastasis, or death from any cause, whichever occur first.

SECONDARY OUTCOMES:
Overall survival | 2 years
  The time from randomization to death from any cause or censored at the date of the last follow-up.
Local-Regional failure free survial | 2 years
  The time from randomization to documented local and/or regional recurrence, or death from any cause.
Distant metastasis-free survival | 2 years
  The time from randomization to distant metastasis or death from any cause.
Complete Response Rate | 9 weeks
  CR is assessed by independent reviewers after induction chemotherapy, according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST v1.1). Complete response is defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) .
  Complete response rate is defined as the percentage of evaluable patients achieving Complete Response following induction chemotherapy.
Incidence of Acute and Late Toxicity | 2 years
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong

IPD SHARING:
Plan to Share IPD: No